CLINICAL TRIAL: NCT03593343
Title: The Effect of Modulating Hepatic Glycogen Content on Hepatic Fat Oxidation
Brief Title: Hepatic Glycogen and Fat Oxidation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL66264.068.18
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Fatty Liver, Nonalcoholic; Meal Time; Fasting; Glycogen Depletion
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fasting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short overnight fast (Experimental): Overnight fasting duration intervention: Participants will receive their last evening meal at 11 pm and stay overnight fasted afterwards for (9.5h).
  Interventions: Behavioral: Overnight fasting duration
- Long overnight fast (Experimental): Overnight fasting duration intervention: Participants will receive their last evening meal at 4.30 pm and stay overnight fasted afterwards for (16h).
  Interventions: Behavioral: Overnight fasting duration

INTERVENTIONS:
Behavioral: Overnight fasting duration — Subjects will adhere to overnight fasting protocol for 6 days

SUMMARY:
Excessive fat in the liver is associated with impairments in metabolic health. Low levels of DNL and high levels of hepatic fat oxidation are considered to be protective.

A decrease in glycogen stores has been causally linked to improved whole body fat oxidation. Also on an organ level, it is suggested that hepatic fat oxidation is stimulated by low hepatic glycogen stores. Next to hepatic fat oxidation, DNL may be influenced by hepatic glycogen stores. Some studies have shown that prolongation of fasting time lowers hepatic glycogen content. It is therefore hypothesized that prolonging fasting time will lower glycogen content and thereby increases fat oxidation and decreases DNL in the liver. To this end, hepatic fat oxidation (plasma marker beta-hydroxybutyrate), de novo lipogenesis, hepatic glycogen content and intrahepatic fat content, will be measured upon a short overnight fast and an extended overnight fast in 13 overweight/obese subjects with hepatic steatosis.

DETAILED DESCRIPTION:
Rationale:

Excessive fat in the liver is associated with impairments in metabolic health. Hepatic lipid storage can originate from several metabolic pathways, including de novo lipogenesis (DNL). On the other hand, there are several metabolic pathways that can decrease hepatic fat storage, such as hepatic fat oxidation. Therefore, low levels of DNL and high levels of hepatic fat oxidation are considered to be protective.

A decrease in glycogen stores has been causally linked to improved whole body fat oxidation. Also on an organ level, it is suggested that hepatic fat oxidation is stimulated by low hepatic glycogen stores. Furthermore, whole body glycogen levels were also linked to DNL and in situations with increased whole body glycogen levels in animal models rates of DNL were also high. Therefore, next to hepatic fat oxidation, DNL may be influenced by hepatic glycogen stores.

Some studies have shown that prolongation of fasting time lowers hepatic glycogen content. It is therefore hypothesized that prolonging fasting time will lower glycogen content and thereby increases fat oxidation and decreases DNL in the liver.

Objective:

The primary objective of this study is to investigate to what extent hepatic fat oxidation can be stimulated by lowering hepatic glycogen content during a prolonged overnight fast.

The secondary objective is to investigate whether reductions in hepatic glycogen content are also accompanied by a decrease in DNL. In addition, the metabolic response to a meal (metabolites related to energy metabolism and substrate oxidation) will be studied upon prolonged overnight fasting. Finally, it will be studied whether reducing hepatic glycogen content by prolonged overnight fasting during a few consecutive days lowers intrahepatic fat storage and changes hepatic fat composition.

Study design:

This is a randomized cross-over study.

Study population:

Thirteen healthy overweight/obese males and postmenopausal females, aged between 45-75 years and BMI between 27-38 kg/m2, with liver fat content ≥ 5% will participate in the study. To be able to include enough people with a liver fat content ≥5%, around 27 participants are expected to be screened for liver fat. When liver fat content is <5%, participants will not be included in the study after determination of liver fat content.

Main study parameters/endpoints:

The primary study outcome is hepatic fat oxidation measured as plasma beta-hydroxybutyrate (BHB) levels, which will be measured before and after one night adherence to the fasting protocols. The secondary study outcome is DNL as determined by stable isotope techniques and will also be measured after one night adherence to the fasting protocols. Other study outcomes include hepatic glycogen content, substrate oxidation and plasma metabolites related to energy metabolism (measured before and after one night adherence to the fasting protocols) and intrahepatic fat content and composition (measured after 6 days of adherence to the fasting protocols).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Caucasian (people will be excluded when having a ≥50% racial African/Asian background)
* Male or postmenopausal female
* Aged 45-75 years at start of the study
* Body mass index (BMI) 27 - 38 kg/m2
* Stable dietary habits (no weight loss or gain >3kg in the past 3 months)
* Sedentary lifestyle (not more than 2 hours of sports per week)
* Liver fat ≥5% as determined by 1H-MRS

Exclusion Criteria:

* Type 2 diabetes
* Active diseases (cardiovascular, diabetes, liver, kidney, cancer or other)
* Contra-indication for MRI (which can be found in appendix II)
* Alcohol consumption of >2 servings per day
* Regular smoking (>5 cigarettes per day)
* No use of medication interfering with investigated study parameters (as determined by responsible physician)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Hepatic fat oxidation | 5 hours
  measured as plasma BHB levels

SECONDARY OUTCOMES:
De novo lipogenesis (DNL) | 20 hours
  measured as percentage of palmitate in VLDL-TG originating from DNL

OTHER OUTCOMES:
Hepatic glycogen content | 1 hour
  Measured with 13C-MRS
Intrahepatic fat accumulation and composition | 20 minutes
  Measured with 1H-MRS
Substrate oxidation | 30 minutes
  measured with indirect calorimetry
Plasma metabolites related to energy metabolism | 5 hours
  measured in plasma samples
Body composition | 5 minutes
  fat mass/fat free mass measured with BodPod

CONTACTS AND LOCATIONS:
Overall Officials: Vera Schrauwen-Hinderling, Dr, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No